CLINICAL TRIAL: NCT04873427
Title: In Situ Clonal Heterogeneity in Prostatic Diagnostic Biopsies: Impact on Prostate Cancer Evolution and Clinical Outcome. A Retrospective, Proof of Concept Study
Brief Title: In Situ Clonal Heterogeneity in Prostatic Diagnostic Biopsies
Status: Terminated | Type: Observational
Why Stopped: The results of the genomic analyses were compromised due to the low DNA concentration.
Sponsor: Clinica Luganese Moncucco (Other)
Responsible Party: Principal Investigator, Marco Roncador, Principal Investigator, Clinica Luganese Moncucco
Other Study IDs: CLM_RAD_001
Record Dates: First submitted 2021-04-28; First posted 2021-05-05 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Prostate Cancer; Genetic Predisposition
Keywords: Prostate Cancer; genetic heterogeneity; personalized medicine
MeSH Terms: conditions — Prostatic Neoplasms; Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — prostatic diagnostic biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- early metastatic prostate cancer patients: Reconstruction of local PCa heterogeneity in multi-needle diagnostic biopsy with different Gleason scores (6-10) using high-coverage whole exome sequencing (WES) and DP-based clonal analysis
  Interventions: Genetic: clonal heterogeneity evaluation
- non-relapsing/non-metastatic patients with indolent malignant disease: Reconstruction of local PCa heterogeneity in multi-needle diagnostic biopsy with different Gleason scores (6-10) using high-coverage whole exome sequencing (WES) and DP-based clonal analysis
  Interventions: Genetic: clonal heterogeneity evaluation

INTERVENTIONS:
Genetic: clonal heterogeneity evaluation — Reconstruction of local PCa heterogeneity in multi-needle diagnostic biopsy with different Gleason scores (6-10) using high-coverage whole exome sequencing (WES) and DP-based clonal analysis

SUMMARY:
This is a retrospective, proof of concept study, which aims at reconstructing the cellular heterogeneity of the tumor in multi-needle diagnostic prostate biopsy as well as any biopsy containing potentially pre-malignant tissue, to study its implications in the clinical history of the disease. For each patient, 2 or more samples will be prepared starting from the FFPE diagnostic material. The biopsy used for assigning the Gleason score will be sequenced, together with two or more of the local peri-proximal biopsies with a higher level of differentiation. Samples will undergo Whole Exome Sequencing with an average coverage of 300x at the Wellcome Sanger Institute (WSI, Hinxton, UK). Sequencing data will be analysed for single nucleotide variants, copy number variants and structural variants by using state-of-the-art data analysis pipeline at WSI.

1. Reconstruction of local PCa heterogeneity in multi-needle diagnostic biopsy with different Gleason scores (6-10) using high-coverage whole exome sequencing (WES) and DP-based clonal analysis;
2. Characterization of the relationships between pathological differentiation (Gleason score) and genomics-measured heterogeneity and malignancy features;
3. Assessment of clinical implications of clonal heterogeneity.

The study will include an average of 150 prostatic diagnostic biopsies from a cohort of 20 early metastatic PC patients and 20 non-relapsing/non-metastatic patients with indolent malignant disease.

DETAILED DESCRIPTION:
Prostate cancer (PCa) is the leading malignancy of the male population. In current clinical practice, diagnostic confirmation of PCa is based on image-guided multi-needle biopsy, in order to capture the intrinsic biological heterogeneity of tumors and to provide a more accurate prediction of clinical outcomes. However, current morphology-based approaches (Gleason score) may not completely describe the complexity of a malignant gland. Not enough is currently known on the impact of genomic heterogeneity in a poorly-differentiated prostate, especially with regards to the development of an indolent versus metastatic prostate malignancy

This is a retrospective, proof of concept study, which aims at reconstructing the cellular heterogeneity of the tumor in multi-needle diagnostic prostate biopsy as well as any biopsy containing potentially pre-malignant tissue, to study its implications in the clinical history of the disease. For each patient, 2 or more samples will be prepared starting from the FFPE diagnostic material. The biopsy used for assigning the Gleason score will be sequenced, together with two or more of the local peri-proximal biopsies with a higher level of differentiation. Samples will undergo Whole Exome Sequencing with an average coverage of 300x at the Wellcome Sanger Institute (WSI, Hinxton, UK). Sequencing data will be analysed for single nucleotide variants, copy number variants and structural variants by using state-of-the-art data analysis pipeline at WSI.

1. Reconstruction of local PCa heterogeneity in multi-needle diagnostic biopsy with different Gleason scores (6-10) using high-coverage whole exome sequencing (WES) and DP-based clonal analysis;
2. Characterization of the relationships between pathological differentiation (Gleason score) and genomics-measured heterogeneity and malignancy features;
3. Assessment of clinical implications of clonal heterogeneity.

The study will include an average of 150 prostatic diagnostic biopsies from a cohort of 20 early metastatic PC patients and 20 non-relapsing/non-metastatic patients with indolent malignant disease.

Descriptive statistics will be carried out and a Mann-Whitney test will be applied on a synthetic parameter for each patient biopsy heterogeneity result, grouped by indolent vs aggressive disease cohort.

The null hypotheses (no difference between the two cohort in heterogeneity) will be rejected if p < 0.05.

The proposed project will evaluate the impact of diagnostic intra-prostatic cell heterogeneity on the clinical course of PCa. The potential prognostic value of local disease clonality could indeed impact the clinical practice: patient with Gleason <7 and lower level of clonal heterogeneity may be moved from an active disease treatment to an active surveillance (AS) approach, avoiding overtreatment for the subjects. Conversely, patients with a similar Gleason score but a more heterogenous malignant population may be required to undergo more aggressive procedures.

ELIGIBILITY:
The inclusion criteria for the subjects in the indolent cohort will be:

* a local disease with Gleason ≤ 7 (3+4, i.e. more differentiated tissue is found in diagnostic biopsies, better overall prognosis)
* no metastasis whatsoever during the follow-up;

The inclusion criteria in the early-metastatic aggressive cohort will be:

* an advanced prostatic neoplasia with Gleason score ≥ 7 (4+3, i.e. less differentiated tissue is found in diagnostic biopsies, worse overall prognosis)
* multiple synchronous or metachronous metastasis.

Exclusion Criteria:

* insufficient material on the tissue biopsy to be left in archives for further evaluations/analyses;
* insufficient amount of tumor cells at baseline;

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — male as we are investigated prostate cancer
Study Population: patients with prostate cancer
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
reconstruction of local PCa heterogeneity | through study completion, an average of 2 years
  Primary endpoint is the reconstruction of local PCa heterogeneity in multi-needle diagnostic biopsy with different Gleason scores (6-10) using high-coverage whole exome sequencing (WES) and DP-based clonal analysis

SECONDARY OUTCOMES:
relationships between pathological differentiation (Gleason score) and genomics-measured heterogeneity | through study completion, an average of 2 years
  Secondary endpoints are characterization of the relationships between pathological differentiation (Gleason score) and genomics-measured heterogeneity and malignancy features; and assessment of clinical implications of clonal heterogeneity.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Franzetti Pellanda, MD, Principal Investigator — Clinica Luganese Moncucco
Locations (1):
- Alessandra Franzetti Pellanda, Lugano, Canton Ticino, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Altmann A, Weber P, Bader D, Preuss M, Binder EB, Muller-Myhsok B. A beginners guide to SNP calling from high-throughput DNA-sequencing data. Hum Genet. 2012 Oct;131(10):1541-54. doi: 10.1007/s00439-012-1213-z. Epub 2012 Aug 11. PMID 22886560
- [Background] Beltran H, Prandi D, Mosquera JM, Benelli M, Puca L, Cyrta J, Marotz C, Giannopoulou E, Chakravarthi BV, Varambally S, Tomlins SA, Nanus DM, Tagawa ST, Van Allen EM, Elemento O, Sboner A, Garraway LA, Rubin MA, Demichelis F. Divergent clonal evolution of castration-resistant neuroendocrine prostate cancer. Nat Med. 2016 Mar;22(3):298-305. doi: 10.1038/nm.4045. Epub 2016 Feb 8. PMID 26855148
- [Background] Bolger AM, Lohse M, Usadel B. Trimmomatic: a flexible trimmer for Illumina sequence data. Bioinformatics. 2014 Aug 1;30(15):2114-20. doi: 10.1093/bioinformatics/btu170. Epub 2014 Apr 1. PMID 24695404
- [Background] Bolli N, Avet-Loiseau H, Wedge DC, Van Loo P, Alexandrov LB, Martincorena I, Dawson KJ, Iorio F, Nik-Zainal S, Bignell GR, Hinton JW, Li Y, Tubio JM, McLaren S, O' Meara S, Butler AP, Teague JW, Mudie L, Anderson E, Rashid N, Tai YT, Shammas MA, Sperling AS, Fulciniti M, Richardson PG, Parmigiani G, Magrangeas F, Minvielle S, Moreau P, Attal M, Facon T, Futreal PA, Anderson KC, Campbell PJ, Munshi NC. Heterogeneity of genomic evolution and mutational profiles in multiple myeloma. Nat Commun. 2014;5:2997. doi: 10.1038/ncomms3997. PMID 24429703
- [Background] Chen X, Schulz-Trieglaff O, Shaw R, Barnes B, Schlesinger F, Kallberg M, Cox AJ, Kruglyak S, Saunders CT. Manta: rapid detection of structural variants and indels for germline and cancer sequencing applications. Bioinformatics. 2016 Apr 15;32(8):1220-2. doi: 10.1093/bioinformatics/btv710. Epub 2015 Dec 8. PMID 26647377
- [Background] Cibulskis K, Lawrence MS, Carter SL, Sivachenko A, Jaffe D, Sougnez C, Gabriel S, Meyerson M, Lander ES, Getz G. Sensitive detection of somatic point mutations in impure and heterogeneous cancer samples. Nat Biotechnol. 2013 Mar;31(3):213-9. doi: 10.1038/nbt.2514. Epub 2013 Feb 10. PMID 23396013
- [Background] Epstein JI, Allsbrook WC Jr, Amin MB, Egevad LL; ISUP Grading Committee. The 2005 International Society of Urological Pathology (ISUP) Consensus Conference on Gleason Grading of Prostatic Carcinoma. Am J Surg Pathol. 2005 Sep;29(9):1228-42. doi: 10.1097/01.pas.0000173646.99337.b1. No abstract available. PMID 16096414
- [Background] Epstein JI, Zelefsky MJ, Sjoberg DD, Nelson JB, Egevad L, Magi-Galluzzi C, Vickers AJ, Parwani AV, Reuter VE, Fine SW, Eastham JA, Wiklund P, Han M, Reddy CA, Ciezki JP, Nyberg T, Klein EA. A Contemporary Prostate Cancer Grading System: A Validated Alternative to the Gleason Score. Eur Urol. 2016 Mar;69(3):428-35. doi: 10.1016/j.eururo.2015.06.046. Epub 2015 Jul 10. PMID 26166626
- [Background] Ferguson, T. S., 1973. A Bayesian analysis of some nonparametric problems.. Annals of Statistics, Volume 1, pp. 209-230.
- [Background] Gandellini P, Casiraghi N, Rancati T, Benelli M, Doldi V, Romanel A, Colecchia M, Marenghi C, Valdagni R, Demichelis F, Zaffaroni N. Core Biopsies from Prostate Cancer Patients in Active Surveillance Protocols Harbor PTEN and MYC Alterations. Eur Urol Oncol. 2019 May;2(3):277-285. doi: 10.1016/j.euo.2018.08.010. Epub 2018 Sep 10. PMID 31200842
- [Background] Hamid AA, Gray KP, Shaw G, MacConaill LE, Evan C, Bernard B, Loda M, Corcoran NM, Van Allen EM, Choudhury AD, Sweeney CJ. Compound Genomic Alterations of TP53, PTEN, and RB1 Tumor Suppressors in Localized and Metastatic Prostate Cancer. Eur Urol. 2019 Jul;76(1):89-97. doi: 10.1016/j.eururo.2018.11.045. Epub 2018 Dec 12. PMID 30553611
- [Background] Helpap B, Egevad L. Modified Gleason grading. An updated review. Histol Histopathol. 2009 May;24(5):661-6. doi: 10.14670/HH-24.661. PMID 19283673
- [Background] Hofman MS, Emmett L. Tumour Heterogeneity and Resistance to Therapy in Prostate Cancer: A Fundamental Limitation of Prostate-specific Membrane Antigen Theranostics or a Key Strength? Eur Urol. 2019 Oct;76(4):479-481. doi: 10.1016/j.eururo.2019.07.030. Epub 2019 Jul 25. No abstract available. PMID 31351666
- [Background] Hugosson J, Carlsson S. Overdetection in screening for prostate cancer. Curr Opin Urol. 2014 May;24(3):256-63. doi: 10.1097/MOU.0000000000000054. PMID 24670870
- [Background] Li H, Durbin R. Fast and accurate short read alignment with Burrows-Wheeler transform. Bioinformatics. 2009 Jul 15;25(14):1754-60. doi: 10.1093/bioinformatics/btp324. Epub 2009 May 18. PMID 19451168
- [Background] Maura F, Bolli N, Angelopoulos N, Dawson KJ, Leongamornlert D, Martincorena I, Mitchell TJ, Fullam A, Gonzalez S, Szalat R, Abascal F, Rodriguez-Martin B, Samur MK, Glodzik D, Roncador M, Fulciniti M, Tai YT, Minvielle S, Magrangeas F, Moreau P, Corradini P, Anderson KC, Tubio JMC, Wedge DC, Gerstung M, Avet-Loiseau H, Munshi N, Campbell PJ. Genomic landscape and chronological reconstruction of driver events in multiple myeloma. Nat Commun. 2019 Aug 23;10(1):3835. doi: 10.1038/s41467-019-11680-1. PMID 31444325
- [Background] Middleton LW, Shen Z, Varma S, Pollack AS, Gong X, Zhu S, Zhu C, Foley JW, Vennam S, Sweeney RT, Tu K, Biscocho J, Eminaga O, Nolley R, Tibshirani R, Brooks JD, West RB, Pollack JR. Genomic analysis of benign prostatic hyperplasia implicates cellular re-landscaping in disease pathogenesis. JCI Insight. 2019 May 16;5(12):e129749. doi: 10.1172/jci.insight.129749. PMID 31094703
- [Background] Nik-Zainal S, Alexandrov LB, Wedge DC, Van Loo P, Greenman CD, Raine K, Jones D, Hinton J, Marshall J, Stebbings LA, Menzies A, Martin S, Leung K, Chen L, Leroy C, Ramakrishna M, Rance R, Lau KW, Mudie LJ, Varela I, McBride DJ, Bignell GR, Cooke SL, Shlien A, Gamble J, Whitmore I, Maddison M, Tarpey PS, Davies HR, Papaemmanuil E, Stephens PJ, McLaren S, Butler AP, Teague JW, Jonsson G, Garber JE, Silver D, Miron P, Fatima A, Boyault S, Langerod A, Tutt A, Martens JW, Aparicio SA, Borg A, Salomon AV, Thomas G, Borresen-Dale AL, Richardson AL, Neuberger MS, Futreal PA, Campbell PJ, Stratton MR; Breast Cancer Working Group of the International Cancer Genome Consortium. Mutational processes molding the genomes of 21 breast cancers. Cell. 2012 May 25;149(5):979-93. doi: 10.1016/j.cell.2012.04.024. Epub 2012 May 17. PMID 22608084
- [Background] Nik-Zainal S, Van Loo P, Wedge DC, Alexandrov LB, Greenman CD, Lau KW, Raine K, Jones D, Marshall J, Ramakrishna M, Shlien A, Cooke SL, Hinton J, Menzies A, Stebbings LA, Leroy C, Jia M, Rance R, Mudie LJ, Gamble SJ, Stephens PJ, McLaren S, Tarpey PS, Papaemmanuil E, Davies HR, Varela I, McBride DJ, Bignell GR, Leung K, Butler AP, Teague JW, Martin S, Jonsson G, Mariani O, Boyault S, Miron P, Fatima A, Langerod A, Aparicio SA, Tutt A, Sieuwerts AM, Borg A, Thomas G, Salomon AV, Richardson AL, Borresen-Dale AL, Futreal PA, Stratton MR, Campbell PJ; Breast Cancer Working Group of the International Cancer Genome Consortium. The life history of 21 breast cancers. Cell. 2012 May 25;149(5):994-1007. doi: 10.1016/j.cell.2012.04.023. Epub 2012 May 17. PMID 22608083
- [Background] Pernar CH, Ebot EM, Wilson KM, Mucci LA. The Epidemiology of Prostate Cancer. Cold Spring Harb Perspect Med. 2018 Dec 3;8(12):a030361. doi: 10.1101/cshperspect.a030361. PMID 29311132
- [Background] Pietzak EJ, Resnick MJ, Mucksavage P, Van Arsdalen K, Wein AJ, Malkowicz SB, Guzzo TJ. Multiple repeat prostate biopsies and the detection of clinically insignificant cancer in men with large prostates. Urology. 2014 Aug;84(2):380-5. doi: 10.1016/j.urology.2014.04.029. Epub 2014 Jun 12. PMID 24929944
- [Background] Shen R, Seshan VE. FACETS: allele-specific copy number and clonal heterogeneity analysis tool for high-throughput DNA sequencing. Nucleic Acids Res. 2016 Sep 19;44(16):e131. doi: 10.1093/nar/gkw520. Epub 2016 Jun 7. PMID 27270079
- [Background] Sved PD, Gomez P, Manoharan M, Kim SS, Soloway MS. Limitations of biopsy Gleason grade: implications for counseling patients with biopsy Gleason score 6 prostate cancer. J Urol. 2004 Jul;172(1):98-102. doi: 10.1097/01.ju.0000132135.18093.d6. PMID 15201746